CLINICAL TRIAL: NCT06264349
Title: Women and Maternity: Development of a Nutritional Education Project
Acronym: MATER
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pavia (Other)
Responsible Party: Principal Investigator, Hellas Cena, Professor, University of Pavia
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 05102023
Record Dates: First submitted 2023-10-05; First posted 2024-02-16 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Pregnancy; Lactation
Keywords: Lifestyle; Health; First one-thousand days; Dietary habits
MeSH Terms: conditions — Breast Feeding; Feeding Behavior

STUDY DESIGN:
Intervention Model Description: Quasi-experimental - controlled, non-randomized pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A: frontal lessons (Experimental): 50 women will receive a Lifestyle Educational Intervention (LEI) from research staff regarding a correct lifestyle during pregnancy and lactation through 6 interactive online lectures lasting approximately 30 minutes each.
  Interventions: Other: Lifestyle Educational Intervention
- Group B: web-mobile app (Experimental): 50 women will receive Lifestyle Educational Intervention (LEI) from research staff regarding a correct lifestyle during pregnancy and lactation through a digital tool (web-mobile app), previously developed.
  Interventions: Other: Lifestyle Educational Intervention
- Control Group (No Intervention): 50 women of the same age as the intervention group will be selected within the LIfestyle and Microbiome InTeraction) Early Adiposity Rebound in Children (LIMIT) project cohort. The LIMIT protocol is registered on clinicaltrials.gov (NCT04960670)

INTERVENTIONS:
Other: Lifestyle Educational Intervention — The Lifestyle Educational Intervention (LEI) consists of promoting a healthy lifestyle during pregnancy and breastfeeding. In particular, the contents concern: i). macro- and micronutrient requirements during pregnancy/breastfeeding; ii). definition of the concept of the food pyramid and healthy plate also considering aspects of food sustainability; iii). definition of the principles of food safety during pregnancy; iv). importance of maternal and infant sleep quality; v). importance of maternal physical activity during pregnancy and lactation; vi). psychological aspects regarding the mother-child dyad.
  Other Names: LEI
  Arms: Group A: frontal lessons; Group B: web-mobile app

SUMMARY:
The "first 1000 days of life", from conception to 2 years of life, are crucial for promoting the health of both mother and baby. During this period, a woman's diet and lifestyle play a significant role in determining the future health of the child. The perinatal period is an ideal time for regular contact with healthcare providers who can institute an intervention to encourage pregnant women to make nutritional changes to improve their health and that of their babies.

Therefore, an educational program on an appropriate lifestyle during the "first 1000 days" can represent a crucial primary prevention strategy in reducing the risk of developing obesity and non-communicable diseases (NCDs) during childhood and later adulthood.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years;
* first trimester;
* parents' ability to speak and understand the Italian language;
* parents' ability to sign the informed consent and to fill in the questionnaires

Exclusion criteria:

* age < 18 years;
* diagnosis of chronic and/or eating disorders

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant women (first trimester)
Enrollment: 100 (Estimated)
Dates: Start 2024-03-15 (Estimated); Primary Completion 2025-05-15 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Gestational weight gain management | GWG will be evaluated at T2 (1 month after delivery)
  Evaluation of the LEI program effectiveness on gestational weight gain (GWG) management. GWG (Kg) will be calculated retrospectively as the difference between the weight at the first and last prenatal visit, just before delivery. Based on that, women will be classified into 3 categories, according to the IOM (U.S.) and the National Research Council (U.S.) Committee to Reexamine IOM Pregnancy Weight Guidelines, as follow:
  i.) Women with Adequate GWG (AGWG; women with normal pre-pregnancy BMI, gaining from 11.5 Kg to 16 Kg during pregnancy); ii.) Women with Excessive GWG (EGWG; women with pre-pregnancy BMI indicating overweight or obesity, gaining more than 11.5 Kg or 9 Kg during pregnancy, respectively); and iii.)Women with Low GWG (LGWG; women with low pre-pregnancy weight status, gaining less than 12.5 Kg).

SECONDARY OUTCOMES:
Nutritional aspects evaluation during pregnancy and lactation | Nutritional aspects will be evaluated at the baseline (T0, first trimester) and after the LEI intervention (T1, three weeks before the delivery; T2, 4 weeks after the delivery; T3, 24 weeks after the delivery).
  Evaluation of the LEI program effectiveness on nutritional aspects. In particular, maternal adherence to the Mediterranean Diet as well as maternal nutritional knowledge will be assessed by meaning of previously validated questionnaires at the baseline (T0, first trimester) and after the LEI intervention (T1, three weeks before the delivery; T2, 4 weeks after the delivery; T3, 24 weeks after the delivery).
Physical activity evaluation during pregnancy and lactation | Physical activity will be evaluated at the baseline (T0, first trimester) and after the LEI intervention (T1, three weeks before the delivery; T2, 4 weeks after the delivery; T3, 24 weeks after the delivery).
  Evaluation of the LEI program effectiveness on physical activity. In particular, to investigate physical activity patterns, a section of a previously developed and validated questionnaire on an Italian youth population was adapted and administered to our adult participants by deleting physical activities in the school environment. This adapted version was also pre-tested on a sample of 24 subjects and revised accordingly. All answers were structured to quantify the time spent weekly in physical activity, including the activities spent during free time and screen time. The questionnaire was composed of 5 multiple-choice questions that followed a Likert scale format comprising 4 choices ("Always", "Often", "Sometimes", and "Never") corresponding to a score between 0 to 3, where the highest score suggested the healthiest habit.
Smoking habits during pregnancy and lactation | Smoking habits will be evaluated at the baseline (T0, first trimester) and after the LEI intervention (T1, three weeks before the delivery; T2, 4 weeks after the delivery; T3, 24 weeks after the delivery).
  Evaluation of the LEI program effectiveness on smoking habits. In particular, smoking habits will be monitored through interviews, and the number of smoked cigarette packs per year will be documented. Participants will be categorized as those who had never smoked, quit smoking before or during pregnancy, or started or kept smoking during pregnancy and/or lactation.
Maternal attitude towards infant feeding. | Maternal attitude towards infant feeding will be evaluated at the baseline (T0, first trimester) and after the LEI intervention (T2, 4 weeks after the delivery).
  The Iowa Infant Feeding Attitude Scale (IIFAS) was used to assess the maternal attitude towards infant feeding methods and to predict breastfeeding intention and exclusivity. In brief, the IIFAS is a standardized interview questionnaire on participants' characteristics and habits (age, residence, education, self-assessed socioeconomic status, relationship status, work before pregnancy, back to work after maternity leave, mode of delivery, parity, way of feeding previous babies, planned way of feeding this newborn)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Project funded by the National Recovery and Resilience Plan (NRRP), ONFOOD Research Project, Spoke 5 - Lifelong and Nutrition. — https://onfoods.it/